CLINICAL TRIAL: NCT00381355
Title: Does the Use of a New Written Action Plan Increase Short-term Adherence to Prescribed Medication and Asthma Control in Children Treated for an Asthma Attack in the Emergency Department: A Randomized Controlled Trial.
Brief Title: RCT of a Written Action Plan vs. Usual Care in Children With Acute Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Francine Ducharme, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 051703
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: asthma; children; written action plan; education; guided self-management; efficacy; compliance; b2-agonists; inhaled corticosteroids; oral steroids; relapse; randomised controlled trial; emergency department
MeSH Terms: conditions — Asthma; Patient Compliance; Recurrence; Emergencies

INTERVENTIONS:
Procedure: Written Action Plan for Acute Asthma

SUMMARY:
The objective of the proposed large, high-intensity, randomised controlled trial is to evaluate the real-life effectiveness of providing a written action plan to asthmatic children discharged from the emergency department (ED) or hospital on the short-term adherence to written recommendations (including medication, attendance to asthma education and medical follow-up). main outcome is adherence to prescribed inhaled preventive medication measured by an electronic counter. Secondary outcomes include attendance to asthma education and to medical follow-up, serving by pharmacy of prescription of oral steroids, as well as asthma control measured by questionnaire (Asthma Quiz for Kidz),2 use of rescue ß2-agonists, relapse to emergency room.

DETAILED DESCRIPTION:
The objective of the proposed large, high-intensity, randomised controlled trial is to evaluate the real-life effectiveness of providing a written action plan to asthmatic children discharged from the emergency department (ED) or hospital on the short-term adherence to written recommendations (including medication, attendance to asthma education and medical follow-up). Contrary to the traditional definition of a written action plan,1 i.e., a set of written instructions to follow in case of an exacerbation, we propose to test a new written action plan based on the innovative concept that emphasises the key elements associated with good asthma care: (1) use of preventive medication, (2) need for asthma education, (3) need for regular medical review, (4) environmental control and (5) instructions for use of rescue medication. The main outcome is adherence to prescribed inhaled preventive medication measured by an electronic counter. Secondary outcomes include attendance to asthma education and to medical follow-up, serving by pharmacy of prescription of oral steroids, as well as asthma control measured by questionnaire (Asthma Quiz for Kidz),2 use of rescue ß2-agonists, relapse to emergency room. Because of the recommended medical follow-up where primary care physicians may recommend a change in the preventive treatment initiated in hospital, only short-term outcomes occurring within 28 days of the index visit will be considered as associated with the use of the written action plan. We have purposely designed this trial to test the additional benefit of the intervention over the usual care, recognizing the heterogeneity in the amount of asthma information provided within the time constraints of the emergency room by our 90 physicians. To provide clinically meaningful and generalisable information, the eligibility criteria for study entry have been limited to the bare necessity to confirm the diagnosis of asthma. The randomisation will be stratified on age to reflect the target interlocutor of the written action plan, namely the parents for the 60% children aged < 6 years, the child and parent pair for the 40% children aged 7 to 12 years old, and the adolescents for the 10% patients aged 13-17 years old. We anticipate important variations in the characteristics of enrolled patients reflecting the real heterogeneity of the emergency department attendees, namely in the severity of baseline exacerbation (55% mild, 35% moderate, 10% severe), ownership of a written action plan (15%), prior asthma education (30%), use of daily preventive medicine (25%), etc, all of which may influence the adherence rate to the written action plan. To compensate this heterogeneity in patients' characteristics and provided instructions, the power of the trial to identify a clinically important difference in the main outcome has been set at 90% rather than the traditional 80%. The strength of the proposed study is clearly the assessment the real-life effectiveness of providing a new concept written action plan to a high-risk population to improve the main obstacles to good asthma control, namely adherence to preventive medication and attendance to asthma education and regular review.

ELIGIBILITY:
Inclusion Criteria:

Children will be eligible, whether they are discharged from the ED or following a hospital admission, if:

1. aged 1 to 17 years;
2. presenting with acute asthma as per the 2003 Canadian Consensus Statement - The ED physician will be responsible for confirming the diagnosis of asthma;
3. requiring at least one nebulisation of salbutamol;
4. the ED physician plans on prescribing the patient inhaled steroids and/or inhaled b2-agonists delivered by metered dose inhaler or continuing a previously prescribed inhaled steroid;
5. the patient intends to stay in the Province of Quebec in the next 45 days;
6. the patient (and their parents) have a good understanding of written and spoken French or English.

Exclusion Criteria:

Children will be excluded if they:

1. currently take asthma medications (ß2-agonist and/or inhaled steroids) using a turbuhaler or diskus, because these delivery devices cannot be fitted with Doser CT, a computerized electronic dose counter for metered dose inhalers;
2. have another chronic lung disease (other than asthma) such as cystic fibrosis or bronchopulmonary dysplasia;
3. have known hypersensitivity to inhaled salbutamol or fluticasone.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Adherence rate to daily inhaled steroids, reported as the ratio of the sum of number of recorded over prescribed activation per day during the 28 days following the index visit.

SECONDARY OUTCOMES:
Proportion of children filling their prescription of oral steroids
Use of rescue B2-agonists measured by dose counter
Quality of life in children aged 7 years and older, measured by the Juniper Questionnaire
Quality of life of their parent, measured by the Juniper Questionnaire
Asthma control, measured by the Asthma Quiz for Kidz
Attendance to asthma education
Attendance to regular medical review
Return visit rate to the ED

CONTACTS AND LOCATIONS:
Overall Officials: Francine M. Ducharme, MD, MSc, Principal Investigator — CHUS-Ste Justine Hospital
Locations (1):
- Ste-Justine Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ducharme FM, Zemek RL, Chalut D, McGillivray D, Noya FJ, Resendes S, Khomenko L, Rouleau R, Zhang X. Written action plan in pediatric emergency room improves asthma prescribing, adherence, and control. Am J Respir Crit Care Med. 2011 Jan 15;183(2):195-203. doi: 10.1164/rccm.201001-0115OC. Epub 2010 Aug 27. PMID 20802165